CLINICAL TRIAL: NCT04767815
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics and Safety After Oral DWN12088 Administration in Healthy Adult Volunteers
Brief Title: To Evaluate Food Effect on the PK and Safety After Oral DWN12088 Administration in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWN12088102
Record Dates: First submitted 2021-02-15; First posted 2021-02-23 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): * Period 1: A (Fasting)
  * Period 2: B (30 minutes after a High-fat meal)
  * Period 3: C (2 hours after a High-fat meal)
  Interventions: Drug: Diet A group; Drug: Diet B group; Drug: Diet C group
- Sequence 2 (Experimental): * Period 1: B (30 minutes after a High-fat meal)
  * Period 2: C (2 hours after a High-fat meal)
  * Period 3: A (Fasting)
  Interventions: Drug: Diet A group; Drug: Diet B group; Drug: Diet C group
- Sequence 3 (Experimental): * Period 1: C (2 hours after a High-fat meal)
  * Period 2: A (Fasting)
  * Period 3: B (30 minutes after a High-fat meal)
  Interventions: Drug: Diet A group; Drug: Diet B group; Drug: Diet C group
- Sequence 4 (Experimental): * Period 1: A (Fasting)
  * Period 2: C (2 hours after a High-fat meal)
  * Period 3: B (30 minutes after a High-fat meal)
  Interventions: Drug: Diet A group; Drug: Diet B group; Drug: Diet C group
- Sequence 5 (Experimental): * Period 1: C (2 hours after a High-fat meal)
  * Period 2: B (30 minutes after a High-fat meal)
  * Period 3: A (Fasting)
  Interventions: Drug: Diet A group; Drug: Diet B group; Drug: Diet C group
- Sequence 6 (Experimental): * Period 1: B (30 minutes after a High-fat meal)
  * Period 2: A (Fasting)
  * Period 3: C (2 hours after a High-fat meal)
  Interventions: Drug: Diet A group; Drug: Diet B group; Drug: Diet C group

INTERVENTIONS:
Drug: Diet A group — Fasting + DWN12088 200 mg
Drug: Diet B group — 30 minutes after a high-fat meal + DWN12088 200 mg
Drug: Diet C group — 2 hours after a high-fat meal + DWN12088 200 mg

SUMMARY:
The pharmacokinetics (PK) and safety of single oral dose of DWN12088 in healthy adults will be compared and assessed on an empty stomach, after high-fat meal, or 2 hours after high-fat meal.

DETAILED DESCRIPTION:
The pharmacokinetics and safety of single oral dose of DWN12088 in healthy adults will be compared and assessed on an empty stomach, after high-fat meal, or 2 hours after high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged ≥ 19 and ≤ 55 years at screening
2. Subjects with body weight ≥ 55.0 kg (male) or ≥ 45.0 kg (female) with a body mass index (BMI) of ≥ 18.0 kg/m2 to < 27.0 kg/m2 at screening test

   ☞ BMI (kg/m2) = Body weight (kg) / {Height (m)}2
3. Subjects who have given written consent on voluntary decision of participation prior to the screening procedure after being fully informed of and completely understanding this study

Exclusion Criteria:

1. Subjects with current or history of clinically significant hematological disorder, tumor, or immunologic, endocrine, psychiatric, neurological, cardiovascular, respiratory, digestive, hepatobiliary, renal, or urinary disorder
2. Subjects with a history of a gastrointestinal disorder (gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc.) or surgery (except for simple appendectomy or hernia surgery) that may affect the safety and PK assessment of the investigational product (IP)
3. Subjects with clinically significant hypersensitivity to any drugs including the ingredient of the IP (DWN12088) or excipients
4. Subjects determined ineligible for meeting the one of the following on the screening tests conducted within 28 days prior to administration of the IP administration

   ① AST or ALT > 1.5 times the upper limit of normal
   * Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2 based on the modification of diet in renal disease (MDRD) formula ③ QTc interval > 450 ms ④ Positive result in serology (hepatitis B tests, hepatitis C tests, human immunodeficiency virus [HIV] tests, syphilis tests) ⑤ Sitting systolic blood pressure > 150 mmHg or < 90 mmHg or sitting diastolic blood pressure > 100 mmHg or < 50 mmHg after resting for more than 3 minutes
5. Subjects with a history of drug abuse or positive result of using abusive drugs in urine drug screening test within 1 year prior to screening
6. Subjects who used any prescription drugs or herbal medicines within 14 days, or any over-the-counter (OTC) drugs including dietary supplements and vitamin supplements within 7 days prior to the first dose of the IP which are judged to impact the study or the subject's safety by the investigator
7. Subjects who participated in another clinical study and received another IP within 180 days before the first dose of the IP
8. Subjects who donated whole blood within 60 days, donated blood components within 30 days, or received blood transfusion within 30 days prior to the first dose of the IP
9. Subjects who consistently consumed excessive amount of caffein or alcohol (caffein > 5 cups/day, alcohol > 210 g/week) or are unable to refrain from caffein or alcohol intake from 3 days before the first dose to the post study visit (PSV)
10. Subjects who are current smokers (may be selected as subjects if they stopped smoking more than 180 days prior to the first dose of the IP) or unable to stop smoking from 180 days prior to the first dose of the IP to the PSV
11. Subjects who used drugs inducing and inhibiting drug-metabolizing enzymes, such as barbital drugs, within 30 days prior to the first dose of the IP
12. Subjects who consumed grapefruit, grapefruit juice, or grapefruit-containing products from 3 days prior to the first hospitalization to the last discharge of period 3, or are unable to refrain from the intake of grapefruit-containing products during this period
13. Subjects who are on or plan to receive CYP2D6 inducing/inhibiting drugs
14. Female subjects who are pregnant or lactating

    ① All female subjects with childbearing potential except for those who are menopausal or surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), who have a positive pregnancy test (serum hCG or urine hCG)
15. Subjects or their spouses or partners who are unable to use medically acceptable appropriate double-method of contraception or medically acceptable contraception throughout the study period and for at least 4 weeks after the last IP administration, and disagreed to refrain from donating sperms during this period

    * Caution: Woman of childbearing potential is defined as a woman who is not surgically sterile or post-menopausal. Women amenorrhoeic for 12 months without an alternative medical cause will be considered as post-menopausal.
    * Medically acceptable methods of contraception ① Use of intrauterine device (except for copper banded coil and hormonal device) for which pregnancy failure rate is proven, by a subject or spouse (or partner) ② Physical and chemical barrier contraception (male/female condom with spermicide, diaphragm, sponge, cervical cap with spermicide, etc.) ③ Surgical sterilization (vasectomy, salpingectomy, tubal ligation, and hysterectomy) of a subject or spouse (or partner)
16. Subjects determined to be ineligible to participate in the study by the investigator due to reasons other than those specified above

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Cmax of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter
AUClast of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter
Adverse events (AEs) such as subjective and objective symptoms | follow-up 26 days after dosing
  To evaluate safety

SECONDARY OUTCOMES:
AUCinf of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter
Tmax of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter
t1/2 of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter
Vd/F of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter
CL/F of DWN12088 and metabolite | Day 1, Day8 and Day15 of 0 hours, 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours
  To evaluate pharmacokinetics parameter

CONTACTS AND LOCATIONS:
Overall Officials: Jaeseong Oh, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea